CLINICAL TRIAL: NCT02605746
Title: A Phase 0/II Study of Ceritinib (LDK378) in Preoperative Glioblastoma Multiforme (GBM) and CNS Metastasis Patients Scheduled for Resection to Evaluate Central Nervous System (CNS) Penetration
Brief Title: Preoperative Ceritinib (LDK378) in Glioblastoma Multiforme and CNS Metastasis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Novartis (Industry); Wayne State University (Other); Translational Genomics Research Institute (Other)
Responsible Party: Principal Investigator, Nader Sanai, Research Clinician, St. Joseph's Hospital and Medical Center, Phoenix
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PHX15BN068
Record Dates: First submitted 2015-09-08; First posted 2015-11-16 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Glioblastoma; Brain Metastases
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2-4 hours (Experimental): All patients will be orally-administered 10-14 doses of ceritinib 750mg with the final dose occurring at one of three intervals before brain tumor resection. This arm has the last ceritinib dose 2-4 hours prior to craniotomy for tumor resection.
  Interventions: Drug: ceritinib 750mg
- 4-8 hours (Experimental): All patients will be orally-administered 10-14 doses of ceritinib 750mg with the final dose occurring at one of three intervals before brain tumor resection. This arm has the last ceritinib dose 4-8 hours prior to craniotomy for tumor resection.
  Interventions: Drug: ceritinib 750mg
- 22-26 hours (Experimental): All patients will be orally-administered 10-14 doses of ceritinib 750mg with the final dose occurring at one of three intervals before brain tumor resection. This arm has the last ceritinib dose 22-26 hours prior to craniotomy for tumor resection.
  Interventions: Drug: ceritinib 750mg

INTERVENTIONS:
Drug: ceritinib 750mg

SUMMARY:
This is two parallel studies to examine pharmacokinetic (PK), pharmacodynamic (PD), and pharmacogenetic (PG) endpoints following short-interval therapy (10-14) daily doses without dose reduction and interruption) with the ALK (anaplastic lymphoma kinase) small-molecule inhibitor, ceritinib.

The Phase 0 study will investigate:

1. first recurrence GBM patients and
2. patients with CNS metastases from solid tumors such as, but not limited to, NSCLC (non-small cell lung cancer) and melanoma.

The CNS (central nervous system) metastases Phase 0 is designed to identify PK effects (in addition to PD, and PG effects on ALK-positive NSCLC metastases), while the GBM Phase 0 is designed to identify PK, PD, and PG effects in all patients.

DETAILED DESCRIPTION:
This study is being done to learn about a new drug, Ceritinib (LKD378). The results of the study may reveal how the drug works for cancer that spreads to the brain (metastases) and for a type of brain cancer called glioblastoma (GBM). Subjects are persons scheduled to have surgery to remove the tumor.This study would test how much of the new drug is present in the tumor, blood, and cerebrospinal fluid (CSF) after taking the drug orally for 10-14 days before surgery. It is only given to patients who are already scheduled to have surgery to remove a tumor that has returned. If the drug seems to be working for a subject's tumor, subject will have the option to continue to receive it as part of a continuation study looking at the drug effect on preventing the tumor from recurring. Small samples of blood, tumor tissue, and CSF will be taken. These samples will be sent to and analyzed at the Barbara Ann Karmanos Cancer Institute (KCI) and to the Translational Genomics Research Institute (TGen). Subject involvement will be for 10-14 days before surgery and for 30 days following surgery. Patients with ALK+ solid tumors will be provided the option of continuing therapy until tumor progression. ALK positivity will be assessed by approved FISH test (Abbott Molecular Inc) using Vysis break apart probes (defined as 15% or more positive tumor cells), the Ventana IHC (immunohistochemistry) test, and/or NGS (next generation sequencing).

ELIGIBILITY:
Inclusion Criteria:

* One prior resection of GBM or MRI evidence of solid tumor CNS metastasis
* All GBM and NSLC metastases must be ALK+
* Eastern Cooperative Oncology Group performance status ≤2
* Archival tumor tissue block available for research use
* Ability to understand written informed consent
* Recovery from toxicities related to prior anticancer therapies to ≤ grade 2 (CTCAE v 4.03). Exception: patients with any grade alopecia
* The following lab criteria are met:

  * Absolute neutrophil count ≥ 1.5 x 10(9th power)/L
  * Hemoglobin ≥ 8 g/dL
  * Platelets ≥ 75 x 10(9th power)/L
  * Serum total bilirubin ≤ 1.5 x upper limit of normal(ULN), except for patients with Gilbert's syndrome who may be included if total bilirubin ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN
  * Aspartate transaminase (AST) < 3.0 x ULN, except for patients with liver metastasis, who are only included if AST < 5 x ULN; alanine transaminase (ALT) < 3.0 x ULN, except for patients with liver metastasis, who are only included if ALT < 5 x ULN
  * Creatinine clearance ≥ 30 mL/min
* Patient has following lab values or has lab values corrected with supplements to be within normal limits at screening:

  * Potassium ≥ LLN
  * Magnesium ≥ LLN
  * Phosphorus ≥ LLN
  * Total calcium (corrected for serum albumin) ≥ LLN

Exclusion Criteria:

* Co-morbid condition(s) that prevent safe surgical treatment
* Active infection or fever > 38.5°C
* Patients with known hypersensitivity to any excipients of ceritinib
* Prior therapy with ceritinib
* Patients with known history of extensive disseminated bilateral interstitial fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, obliterative bronchiolitis, and clinically significant radiation pneumonitis (affecting activities of daily living or requiring therapeutic intervention)
* Clinically significant uncontrolled heart disease and/or recent cardiac event (within 6 months), such as:

  * history of documented congestive heart failure (New York Heart Association functional classification III-IV);
  * uncontrolled hypertension defined by a Systolic Blood Pressure ≥ 160 mm Hg and/or Diastolic Blood Pressure ≥ 100 mm Hg, with or without antihypertensive medication
  * initiation or adjustment of antihypertensive medication(s) is allowed prior to screening;
  * ventricular arrhythmias; supraventricular and nodal arrhythmias not controlled with medication;
  * other cardiac arrhythmia not controlled with medication;
  * corrected QTc > 450 msec using Fridericia correction on the screening ECG
* Impaired GI function or GI disease that may alter absorption of ceritinib or inability to swallow up to five ceritinib capsules daily
* Ongoing GI adverse events > grade 2 (e.g. nausea, vomiting, or diarrhea) at the start of the study
* Receiving medications that meet 1 of the following criteria and cannot be discontinued at least 1 week prior to start of treatment with ceritinib and for the duration of participation:

  * Medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes
  * Strong inhibitors or strong inducers of CYP3A4/5
  * Medications with a low therapeutic index that are primarily metabolized by CYP3A4/5, CYP2C8 and/or CYP2C9
  * Therapeutic doses of warfarin sodium (Coumadin) or any other coumadin-derived anti-coagulant. Anticoagulants not derived from warfarin are allowed
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential, unless they are using highly effective methods of contraception during dosing and for 3 months after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02-17 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration | at pre-dose on day 10-14(Day 0), 0.5, 1, 2, 4, 6, 8, and 24 hours following single dose of CERITINIB
  Plasma concentration of Ceritinib after 10-14 oral doses of 750 mg. Will be summarized using descriptive statistics.
Cerebrospinal Concentration | collected intraoperatively at 2-4, 4-8, and 22-26 hours following single dose of CERITINIB relative to the final dose on day 10-14
  Cerebrospinal concentration of Ceritinib. Will be summarized using descriptive statistics.
Intratumoral Concentration | collected intraoperatively at 2-4, 4-8, and 22-26 hours following single dose of CERITINIB relative to the final dose on day 10-14
  Intratumoral concentration of Ceritinib. Will be summarized using descriptive statistics.

SECONDARY OUTCOMES:
Tumor Tissue | at baseline(archival) and up to 26 hours post dosing
  Tumor tissue quantification of total and phosphorylated forms of ALK, JAK/STAT5B, and Caspase-3. Will be summarized using descriptive statistics.
Tumor Cells in M-Phase | at baseline and up to 26 hours post dose CERITINIB
  Number of tumor cells in M-phase of cell cycle (PH3). Will be summarized using descriptive statistics.
Double Strand DNA | at baseline and up to 26 hours post dose CERITINIB
  Presence of double-strand DNA damage (γH2AX). Will be summarized using descriptive statistics.
Tissue Concentration | 2-4, 4-8, and 22-26 hours post dosing relative to the final Day 10 dose, as compared to the immediate pre-operative MRI scan
  Tissue concentration of CERITINIB compared to contrast enhancing GBM vs. surrounding nonenhancing FLAIR-hyperintense GBM. Will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Principal Investigator — Barrow Brain and Spine, Phoenix AZ
Locations (1):
- Barrow Brain and Spine, Phoenix, Arizona, United States